CLINICAL TRIAL: NCT04217135
Title: The Prognostic Impact of Using High-dose Hydralazine in Severe Systolic Heart Failure With Hemodynamically Significant Mitral Regurgitation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Shih-Hung Hsiao, Staff of Cardiology, Principal Investigator, Clinical Associate Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EMRP18106N
Record Dates: First submitted 2019-12-29; First posted 2020-01-03 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Systolic Heart Failure Stage D (Disorder); Mitral Regurgitation
Keywords: high-dose hydralazine; mitral regurgitation; severe systolic heart failure; heart failure rehospitalization; all-cause mortality
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure, Systolic | interventions — Hydralazine

STUDY DESIGN:
Intervention Model Description: This prospective study will recruit 400 patients aged 18 years or older, and hospitalization to E-Da Hospital for acute decompensated heart failure due to severe left ventricular systolic dysfunction combined with hemodynamically significant mitral regurgitation. Severe systolic dysfunction and hemodynamically significant mitral regurgitation are defined as left ventricular ejection fraction less than 35% and mitral regurgitant volume more than 45 ml (more than moderate degree), respectively. All participants will be randomly divided into two groups according to 1 to 1 fashion. One group will receive conventional evidence-based medication with up-titration to maximal tolerable dose and another group will receive low-dose hydralazine initially with rapid up-titration, if no adverse effect including hypotension with worsening low cardiac output sign, skin rash and joint pain occurred.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional treatment (Active Comparator): This group will receive conventional evidence-based medications with up-titration to maximal tolerable dose. The evidence-based medications include angiotensin converting enzyme inhibitor/angiotensin receptor blocker, beta-blocker, mineralocorticoid receptor antagonist, ivabradine and entresto. Which evidence-based medications will be started first depends on the decision of in-charge doctors without strict regulation. However, all evidence-based medications should be up-titrated to maximal tolerable dose. (Excuse me! Up-titration of evidence-based medications in heart failure isn't multiple intervention. Those medications should be prescribed in each heart failure case if no contraindication was noted.)
  Interventions: Drug: evidence-based medications vs. high-dose hydralazine + evidence-based medications
- high-dose hydralazine group (Active Comparator): another group will receive low-dose hydralazine initially with rapid up-titration, if no adverse effect including hypotension with worsening low cardiac output sign, skin rash and joint pain occurred. Since the half-life of hydralazine is around 4-6 hours and 3-5 half-life achieves the steady blood concentration, up-titration of hydralazine will be done per 1-2 days. For example, initial dose of hydralazine would be 25 mg tid and the dose would be 50 mg bid next day if no adverse effect occurred. Following this rule, one week is enough to reach high-dose hydralazine with daily dose of 300-400 mg.
  Interventions: Drug: evidence-based medications vs. high-dose hydralazine + evidence-based medications

INTERVENTIONS:
Drug: evidence-based medications vs. high-dose hydralazine + evidence-based medications — randomized in 1 to 1 fashion After discharge, high-dose hydralazine is maintained except any adverse effect and up-titration of other evidence-based medications to maximal tolerable dose will be done. The dose of medications is adjusted by clinical signs, especially peripheral perfusion, not only simply by blood pressure. If participant had low blood pressure (for example, systolic blood pressure less than 90 mmHg) but no sign of postural hypotension, or low cardiac output (cold limbs, decreased urine output, dizzy), the investigators will keep up-titration of medications.

SUMMARY:
Background: Severe systolic heart failure would be complicated with low cardiac output and high left ventricular filling pressure and the clinical presentations would be low blood pressure, poor peripheral perfusion, and pulmonary edema. Severe systolic heart failure with hemodynamically significant mitral regurgitation brings even more challenged since the obvious elevation of left atrial pressure induces more pulmonary congestion and backward flow of regurgitation in cases with already low cardiac output and poor peripheral perfusion complicates more severe of low cardiac output. Surgical interventions in those cases aren't strongly recommended due to very high operation risk. In the era of lack of nitroprusside in Taiwan (more than 7 years), hydralazine, a direct vasodilator, is a potential substitute for treatment of those cases. The advantages of hydralazine include 1) different dosage forms are available (10 mg, 25 mg, and 50 mg); 2) short half-life makes it reaching steady blood concentration in short period and allow to up- titrate rapidly and also recover fast while adverse reaction occurs; 3) it is much cheaper than other evidence-based medications. In this study, the investigators try to use rapid up-titration of hydralazine to maximal tolerable dose, almost up to 300-400 mg per day, combined with other evidence-based medications in cases with left ventricular ejection fraction less than 35% and mitral regurgitation severity more than moderate degree and assess the prognostic impact.

Objective: Four hundred of patients with severe systolic dysfunction and hemodynamically significant mitral regurgitation, who were admitted for intensive care unit for acute decompensated heart failure, will be enrolled and the participants will be divided into two groups according 1 to 1 randomization process. Control group will receive conventional treatment with tolerable maximal dose of evidence-based medications and study group will use hydralazine with rapid up-titration, if no clinical adverse responses were noted, following by or simultaneously using evidence-based medications. The end-points include in- hospital mortality, 3-year all-cause mortality and heart failure rehospitalization.

During follow-up period, any adverse response of high-dose hydralazine including lupus-like syndrome and arthritis will be monitored.

DETAILED DESCRIPTION:
Background:

The investigator team had focused on heart failure (HF) treatment for many years and tried to develop non-invasive guide for HF treatment. Initially, the investigators had dedicated to use echocardiography to simulate Swan-Ganz and performed validation for non-invasive Swan-Ganz (echo Swan-Ganz). Although this method wasn't successful in assessing the full spectrum of Swan-Ganz data, the estimates of stroke volume and left ventricular filling pressure (LVFP) were reliable and well-validated by comparing with invasive measurements. Based on those two data, the investigators could control severe HF patients better and conducted a HF special outpatient clinic. Guiding HF treatment by this model was on-going. Due to lack of nitroprusside in Taiwan for more than 8 years, some cases with terminal HF combined with severe mitral regurgitation or aortic regurgitation were more complicated and troubled for management since it might present as even more reduction of forward flow with more low cardiac output and high LVFP. High-dose of hydralazine, a direct vasodilator, was the solution of our team and it was used to a substitute of nitroprusside. According to the preliminary results of previous studies, rapid up-titration of hydralazine to maximal tolerable dose, then combined with evidence-based medications, was very effective in patients with severe systolic HF and hemodynamically significant mitral regurgitation, especially in acute pulmonary edema with critical and unstable conditions. This method is useful for reducing regurgitation volume and promoting forward flow after afterload reduction and the counterbalance between increasing forward flow and pressure-lowing effect of vasodilator brings stable blood pressure without obvious hypotension or poor peripheral perfusion. Therefore, it increases the possibility of extubation and reduces the in-hospital mortality in those cases. Additionally, the risk of lupus-like syndrome, arthritis, and positive result of ANA are relatively lower than those in The East population. However, the exact short-term and long-term benefits of high-dose hydralazine in Taiwanese with severe systolic HF and significant mitral regurgitation are unknown. The investigators conduct this study to confirm our previous observation.

Introduction Heart failure, either acute or chronic, is a clinical syndrome caused by a structural and/or functional cardiac abnormality, resulting in a reduced cardiac output and/or elevated intracardiac pressures at rest or during stress. This means two major components associated with HF symptoms are inadequate cardiac output and high filling pressure. Although many categories of medications have been approved as therapeutic interventions for HF, including beta-blockers, angiotensin converting enzyme inhibitors (ACEI), angiotensin receptor antagonists (ARB), mineralocorticoid receptor antagonists (MRA), ivabradine, and entresto, the prognosis of HF remains poor, even worse than that of most cancers. Up-titration of evidence-based medications to maximal tolerable dosages has been recommended, but loop diuretics remain the main stream of HF treatment despite lack of evidence of prognostic benefit. In daily practice, diuretics resolve respiratory distress with reduction preload and LVFP, but overdiuresis with postural hypotension, renal function decline and worsening low cardiac output is not uncommon. Decompensated HF with low blood pressure is always difficult to manage, and most evidence-based medications have blood-pressure-lowing effect at initiation of treatment. Many physicians do not up-titrate those medications to maximal dosages for fear of more reduction of blood pressure, which potentially induces adverse events or complications. Therefore, many eligible patients don't reach suggested dosage according to guidelines, which may adversely affect prognosis. It points out a blind spot of HF treatment that relatively low blood pressure would avoid up-titration of evidence-based medications in daily practice of the majority of cardiologists. Regarding severe systolic HF with hemodynamically significant mitral regurgitation (MR), it is an even more complicated situation because regurgitation will bring much lower stroke volume and higher LVFP, which blood pressure becomes low enough to let physicians withdrawing any medications with blood-pressure-lowering effect, including evidence-based medications. The nitroprusside with powerful vasodilating and short-active (rapid conversion after stopping infusion) effects are the solution of this critical situation. Unfortunately, this medication was unavailable for more than 8 years in Taiwan.

Many short-active medications with vasodilator effect such as captopril and hydralazine have potential to be a substitute of nitroprusside in this situation and are suitable for rapid up-titration because short half-life brings to achieve steady blood concentration soon. Compared to hydralazine, captopril decreases the mortality of advanced HF, mainly sudden death, in line with enalpril. But only the form of captopril 25 mg per tab is available in Taiwan and one fourth tab three times per day is the common initial regimen.

Although ACEIs offer strong prognostic benefit in HF and favorable hemodynamic change, it is not so convenient to use in study cohort. Regarding hydralazine, three forms including 10, 25, and 50 mg are available. Animal study reveals that it is effective for treatment of mitral regurgitation with reduction of peripheral vascular resistance and LVFP, and increase of stroke volume and cardiac output. The effect of hydralazine is comparable to nitroprusside with a similar reduction in systemic vascular resistance but a slightly greater increase in cardiac index, with a lesser fall in mean arterial pressure, mean pulmonary arterial pressure, and pulmonary wedge pressure. Hydralazine combined with nitrate had been documented useful in chronic heart failure, especially in African or black population, according to many publications. Based on the hypothesis that initial low-dose hydralazine with rapid up-titration to maximal tolerable dose, following by or simultaneously using other evidence-based medications, in acute HF patients with low-cardiac-output and low-blood-pressure patients due to severe left ventricular systolic dysfunction and hemodynamically significant mitral regurgitation, would bring better outcome compared to conventional treatment, the investigators conduct this study to assess short-term and long-term prognostic change.

Methods Study population: This prospective study will recruit 400 patients aged 18 years or older, and hospitalization to E-Da Hospital for acute decompensated heart failure due to severe left ventricular systolic dysfunction combined with hemodynamically significant mitral regurgitation. Severe systolic dysfunction and hemodynamically significant mitral regurgitation are defined as left ventricular ejection fraction less than 35% and mitral regurgitant volume more than 45 ml (more than moderate degree), respectively. All participants will be randomly divided into two groups according to 1 to 1 fashion. One group will receive conventional evidence-based medication with up-titration to maximal tolerable dose and another group will receive low-dose hydralazine initially with rapid up-titration, if no adverse effect including hypotension with worsening low cardiac output sign, skin rash and joint pain occurred. Since the half-life of hydralazine is around 4-6 hours and 3-5 half-life achieves the steady blood concentration, up-titration of hydralazine will be done per 1-2 days. For example, initial dose of hydralazine would be 25 mg tid and the dose would be 50 mg bid next day if no adverse effect occurred. Following this rule, one week is enough to reach high-dose hydralazine with daily dose of 300-400 mg. According to our prior experience of acute HF control, the most patients could tolerate this dose well with acceptable peripheral perfusion and blood pressure. This process will follow by or simultaneously use evidence-based medications including ACEI/ARB, beta-blocker, and MRA. Exclusion criteria include any history of the following: 1) cancer or other significant co-morbid diseases with expected life span less than 3 years, 2) any sign of inadequate preload such as poor skin turgor, severe thirsty feeling, evidence of gastrointestinal tract bleeding or sepsis, 3) adverse effects of hydralazine, 4) surgical interventions of mitral regurgitation will be done in follow-up period which change the course of native condition, 5) other valvular conditions other than mitral regurgitation with severity more than or equal to moderate degree, particularly mitral stenosis, and aortic regurgitation/stenosis, or 6) lack of written informed consent. Signs of inadequate peripheral perfusion including downhill consciousness level, decreased urine output, and prerenal azotemia will be assessed routinely. Histories of hyperlipidemia, hypertension, diabetes and smoking are recorded. The endpoints for the current study are in-hospital mortality, 3-year HF rehospitalization and 3-year all-cause mortality. All participants will give written informed consent to participate in the study, and the study had been approved by the institutional review board.

Measurement of hemodynamic change after high-dose hydralazine: Thirty patients in each group will be arranged for admission to intensive care unit for severe HF control, and they will receive invasive hemodynamic monitor by Swan-Ganz catheter routinely for 1 week. Hydralazine will be up-titrated to maximal tolerable dose in hydralazine group at first 7 days and the target dose will be 300-400 mg per day. Echocardiographic measurements including stroke volume, left ventricular ejection fraction, left atrial size, mitral regurgitation severity, mitral regurgitant volume, pulmonary artery systolic pressure, tissue Doppler parameters, and left ventricular filling pressure estimated by left atrial expansion index, will be done at day 1 and day 7.

Maintenance of high-dose hydralazine: After discharge, high-dose hydralazine is maintained except any adverse effect and up-titration of other evidence-based medications to maximal tolerable dose will be done. The dose of medications is adjusted by clinical signs, especially peripheral perfusion, not only simply by blood pressure. If participant had low blood pressure (for example, systolic blood pressure less than 90 mmHg) but no sign of postural hypotension, or low cardiac output (cold limbs, decreased urine output, dizzy), the investigators will keep up-titration of medications. Regarding the initial negative inotropic effect of beta blockers, it will be titrated slowly. While any reasons induce postural hypotension, the investigator will reduce the dose of hydralazine first and try to keep the ordinary dose of other evidence-based medications as possible. If participants would admit for recurrent heart failure or other non-cardiovascular problems, ordinary regimen of high-dose hydralazine will be maintained unless low blood pressure combined with low cardiac output occurs.

Monitor adverse effect of high-dose hydralazine: Antinuclear antibody, hematogram and CXR will be checked per 6 months. Signs of lupus-like syndrome, serositis, joint pain, skin rash, liver biochemical and hematological studies will be monitored regularly. For patients with coronary artery disease and ischemic HF, the investigators will take care of any signs of worsening myocardial ischemia if chest pain occurs or HF worsens.

High-dose captopril will replace hydralazine if any adverse effects of high-dose hydralazine are suspected. Echocardiographic measurements: Basic echocardiographic measurements including left ventricular ejection fraction, pulmonary artery systolic pressure, left atrial size, and tissue Doppler imaging will be done. Echocardiography is performed in all patients. The severity of mitral regurgitation will be evaluated quantitatively by regurgitant volume. Heart failure patients are admitted with left ventricular ejection fraction less than 35% and mitral regurgitant volume more than 45 ml will be enrolled if they are willing to participate in. Left atrial volume measurements were calculated using the biplane area-length method immediately before mitral valve opening. In all participants, the left atrial volumes were indexed to the body surface area. The mitral regurgitation volume is calculated as follows: regurgitation volume = (stroke volume of mitral annulus) - (stroke volume of left ventricular outflow tract), where the stroke volumes of the mitral annulus and left ventricular outflow tract were obtained by multiplying the cross-sectional area by the respective time-velocity integral. The mitral regurgitant volumes will be assessed at enrollment, at discharge, and at least once per year during follow-up period. Based on our prior studies, the change of LVFP assessed by left atrial expansion index will be examined during the course of admission.

Biochemical studies and biomarker measurements: Blood samples will be obtained during index hospitalization and per 3 months after discharge. The measurements of B-type natriuretic peptide, anti-nuclear antibodies, renal function, liver function and hematogram will be done regularly.

Follow up: The median follow-up will be 3 years and the end-points will be in-hospital mortality, 3-year HF rehospitalization and 3-year all-cause mortality. Hospitalization for HF is defined as a hospital stay of at least 1 night for treatment of a clinical syndrome with at least two of the following symptoms: paroxysmal nocturnal dyspnea, orthopnea, elevated jugular venous pressure, pulmonary rales, a third heart sound, cardiomegaly on chest radiography, or pulmonary edema on chest radiography. These clinical signs and symptoms might have represented a clear change from the normal clinical state of the patient and might have been accompanied by either failing cardiac output, as determines by peripheral hypoperfusion, or peripheral or pulmonary edema requiring treatment with intravenous diuretics, inotropes, or vasodilators. Supportive documentation of a decreased cardiac index, an increased pulmonary capillary wedge pressure, decreasing oxygen saturation, and end organ hypoperfusion, if available, are included in the adjudication. Follow-up includes medical record reviews and patient interviews. Medical assistants will check medical records once per 3 months. The certification of death is based on death records, death certificates, and hospital medical records.

Statistical analysis: The SPSS software will be used for all statistical analyses. All continuous variables are presented as means ± standard deviation. A p value of < 0.05 is considered statistically significant. Comparisons of clinical characteristics are performed by chi-square analysis for categorical variables. Acute hemodynamic changes after high-dose hydralazine will be assessed and comparisons of Swan-Ganz and echocardiographic data before and after high-dose hydralazine will be performed. Otherwise, comparisons of hemodynamic changes between conventional treatment group and hydralazine will also be done. Kaplan-Meier curve will be performed to assess the cumulative event-free rate according to different treatment strategies. Cox proportional regression analysis of hazard ratio after adjusting significant covariates in univariate analyses will be done. Otherwise, multivariate analysis will be done to identify the independent prognostic indicators of in-hospital, 3-year HF rehospitalization, and 3-year all-cause mortality. ROC curve analysis is also performed to assess the sensitivity and specificity of the cut-off points of covariates for predicting those events. The frequency of adverse effects of high-dose hydralazine, including positive antinuclear antibody, lupus-like syndrome, serositis, arthritis, hematogram change, and worsening myocardial ischemia will be assessed. If the strategy of high-dose hydralazine combined with conventional evidence-based medications was proved to have prognostically beneficial effect, the prognostic impact according to maximal tolerable dose of hydralazine will be analyzed. Additionally, high dose of hydralazine will compress the use of other evidence-based medications and it is assumed that, compared to conventional treatment group, up-titration of those medications becomes difficult in high-dose hydralazine group. The effect of counter-balance between high-dose hydralazine and relatively low doses of ACEI, ARB, beta blocker and MRA will be assessed by multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* acute decompensated heart failure due to severe left ventricular systolic dysfunction combined with hemodynamically significant mitral regurgitation. Severe systolic dysfunction and hemodynamically significant mitral regurgitation are defined as left ventricular ejection fraction less than 35% and mitral regurgitant volume more than 45 ml (more than moderate degree), respectively

Exclusion Criteria:

* cancer or other significant co-morbid diseases with expected life span less than 3 years
* adverse effects of hydralazine
* surgical interventions of mitral regurgitation will be done in follow-up period which change the course of native condition
* other valvular conditions other than mitral regurgitation with severity more than or equal to moderate degree, particularly mitral stenosis, and aortic regurgitation/stenosis
* lack of written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
in-hospital mortality | From date of randomization until the date of in-hospital death at indexed hospitalization, assessed up to 2 months
  death at indexed hospitalization
3-year heart failure (HF) rehospitalization | From date of randomization until the date of first rehospitalization for heart failure or date of death from any cause, whichever came first, assessed up to 156 months
  Hospitalization for HF is defined as a hospital stay of at least 1 night for treatment of a clinical syndrome with at least two of the following symptoms: paroxysmal nocturnal dyspnea, orthopnea, elevated jugular venous pressure, pulmonary rales, a third heart sound, cardiomegaly on chest radiography, or pulmonary edema on chest radiography.
3-year all-cause mortality | From date of randomization until the date of date of death from any cause, assessed up to 156 months
  The certification of death is based on death records, death certificates, and hospital medical records

CONTACTS AND LOCATIONS:
Locations (1):
- E-Da hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No